CLINICAL TRIAL: NCT02622555
Title: Phase 4 Study of Cardiovascular Morbidity and Safety in Women Treated With Mirabegron for Overactive Bladder
Brief Title: Cardiovascular Morbidity During Treatment of Overactive Bladder With B3 Agonists
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helena Kopp Kallner, Consultant obstetrics gynecology,, Karolinska Institutet
Other Study IDs: DSABHT13
Record Dates: First submitted 2013-06-20; First posted 2015-12-04 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mirabegron treatment: Women with overactive bladder syndrome eligible for Mirabegron treatment
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Patients with overactive bladder eligible for drug treatment who fulfill the EMA prescription guidelines receive mirabegron 50 mg extended release once daily according to clinical routine
  Other Names: Betmiga

SUMMARY:
Overactive bladder syndrome complicates life for many women. 60-70% of women report improvement with treatment but the antikolinergic treatment is often limited by the adverse events, for example dry mouth, obstipation and urinary retention. Mirabegron is a b3-adrenoreceptor agonist which induces detrusor relaxation. Earlier studies has demonstrated similar efficacy comparing Mirabegron with antimuscarinics but a significant reduction of adverse events. The aim of the present study is to survey cardiovascular adverse events with Mirabegron treatment in a general population suffering from overactive bladder syndrome.

DETAILED DESCRIPTION:
Overactive bladder syndrome complicates life for many women. For 30 years the dominant treatment of overactive bladder syndrome has been antimuscarinics as first-line pharmacotherapy. 60-70% of women report improvement with treatment but the therapy is limited by the adverse events, for example dry mouth, obstipation and urin retention. In Sweden, prescription of antimuscarinics has increased by 69% during the period of 2000-2007 which implies an increasing desire to seek treatment.

Mirabegron is a b3-adrenoreceptor agonist which induces detrusor relaxation. Earlier studies have demonstrated similar efficacy when comparing Mirabegron with antimuscarinics but a significant reduction of adverse events. Clinical phase I-III trials have registered an increased pulse rate and effects on blood pressure in some patients. The aim of the present study is to survey cardiovascular adverse events with treatment with Mirabegron in the general population suffering from overactive bladder syndrome.

ELIGIBILITY:
Inclusion Criteria

* Overactive bladder syndrome, eligible for Mirabegron treatment

Exclusion Criteria:

* As specified by regulatory authorities for drug prescription

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General population of women with overactive bladder syndrome without strict exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2013-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline and 2 months
  Change in diastolic and systolic blood pressure from baseline to 2 months follow-up

SECONDARY OUTCOMES:
Heart rate changes | baseline and 2 months
  Changes in heart rate from baseline to 2 months follow-up
Changes in cardiac electrophysiology | Baseline and 2 months
  Recorded ECG changes from baseline to 2 months follow-up
Subjective symptomatic outcome (Urinary Distress Iinventory) | Baseline and 2 months
  Self reported questionnaire data (Urinary Distress Iinventory). Scores reflect changes in condition specific symptoms from baseline to 2 months follow-up
Subjective quality of life outcome (Pelvic Floor Impact Questionnaire) | Baseline and 2 months
  Self reported questionnaire data (Pelvic Floor Impact Questionnaire). Scores reflect changes in condition specific quality of life from baseline to 2 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Altman, Ass. prof., Principal Investigator — Karolinska Institutet
Locations (1):
- Daniel Altman, Stockholm, Stockholm County, Sweden